CLINICAL TRIAL: NCT05823207
Title: Effect of Sage Essential Oil Inhalation Aromatherapy on Premenstrual Syndrome and Quality of Life: A Randomized Controlled Study
Brief Title: Effect of Sage Essential Oil Inhalation Aromatherapy on Premenstrual Symptoms and Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cansu Mine Aydin (Other)
Responsible Party: Sponsor-Investigator, Cansu Mine Aydin, research assistant, Kafkas University
Organization: Kafkas University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KAFKAS-SAG-CMAYDIN-001
Record Dates: First submitted 2023-04-08; First posted 2023-04-21 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Premenstrual Syndrome; Anxiety
Keywords: premenstrual syndrome; aromatherapy; students; sage oil
MeSH Terms: conditions — Premenstrual Syndrome; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The first group will be determined as the experimental group that inhales sage essential oil, and the second group will be determined as the control group. 2 group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sage essential oil (Experimental): Sage essential oil is applied twice a day for a total of 6 drops for 5 days in each cycle.
  Interventions: Other: sage essential oil
- control group (No Intervention): No application was made to this group. Personal information form and PMS scale and quality of life scale will be applied to this group at the end of each cycle.

INTERVENTIONS:
Other: sage essential oil — It will be applied 2 times a day, at the same times, at a distance of 30 cm from the nose for 5 minutes with normal breathing and 3 drops of essential oil by placing a tampon. The PMS scale and the quality of life scale are administered to the participants at the end of the 1st, 2nd and 3rd cycles of the menstrual cycle.
  Arms: Sage essential oil

SUMMARY:
The changes (mood changes, lethargy, irritability, etc.) that gradually disappear with the start of the menstrual period in women are called premenstrual syndrome. Anxiety, irritability, poor concentration, depression, mood swings, lethargy, sleep disturbance, breast tenderness, change in appetite, bloating, headache, weight gain, abdominal pain, fatigue, and gastrointestinal symptoms are seen in this syndrome. Safe and effective treatments are needed as these symptoms negatively affect both work and personal lives of women. Some women also turned to therapeutic approaches due to the high side effects of pharmacological treatment. One of these approaches is the aromatherapy method, which is widely used today. Aromatherapy is a therapy aimed at protecting and improving one's physical, mental and psychological health. Traditionally, aromatherapy has been used as one of the non-pharmacological methods for reducing premenstrual symptoms, releasing uterine cramps, and reducing pain and anxiety. Sage oil, with its ester components, regulates the menstrual cycle and hormonal components and alleviates climatic changes and symptoms in menopausal women. It is also recommended to use sage essential oil to reduce uterine tonics and to reduce fluid retention in the premenstrual period. In our country, no study was found in which aromatherapy was performed using sage oil in PMS. It is thought that the study to be conducted in this area will be beneficial in terms of evaluating the effectiveness of a non-pharmacological method in the treatment of PMS.

DETAILED DESCRIPTION:
In premenstrual symptoms, psychotropic drugs, hormone therapy or nonsteroidal anti-inflammatory drugs are used as pharmacological methods. Aromatherapy, which is one of the non-pharmacological methods, is preferred to reduce premenstrual symptoms. Aromatherapy through massage and inhalation is commonly used in nursing interventions. Sage has also been used for various human ailments since ancient times. Sage oil regulates the menstrual cycle and hormonal components and is known to alleviate climatic changes and symptoms in menopausal women. The main goal of nursing practices is to ensure the well-being of the individual, family and society, to maintain care, to organize attempts to protect and improve health, to teach coping methods for healing and rehabilitation in case of illness, and is to increases the quality of life.

From this point of view, studies have shown that aromatherapy has an effect on reducing premenstrual symptoms and increasing quality of life. This research, It is thought that it will both create a resource for nurses and contribute to the formation of the necessary evidence for the application of sage oil in aromatherapy in people with PMS.

ELIGIBILITY:
Inclusion Criteria:

* Getting over 110 points from the PMS scale,
* Experiencing at least five PMS symptoms each month,
* Not having sexual intercourse
* Regular menstruation, (regular menstruation (between 21-35 days) )
* Absence of any chronic disease,
* Not using any method to deal with PMS
* No known allergic reaction to the essential oil to be used,
* Those who are not bothered by the smell of the essential oil to be used and accept the use of sage essential oil
* Not taking Hormone Replacement Therapy
* Women who agreed to participate in the study were included in the study group.

Exclusion Criteria:

* Married
* Allergy,
* Individuals with inconvenient conditions (nausea, dizziness, febrile diseases, high fever, skin or joint inflammation, unknown itching and redness, unknown edema, open wound, cancer, recent operation, intra-abdominal surgery, cyst, appendicitis) ),
* Irregular menstruation,
* Not having regular periods in the last three months,
* Having a psychiatric diagnosis,
* Having any gynecological disease (abnormal uterine bleeding, myoma, ovarian cyst, etc.)
* Using contraceptive drugs,
* Those with olfactory problems (anosmia)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form: | 1 year
  It will take 10-15 minutes for the participants to fill out the questionnaire consisting of 33. Students who accept the scent of sage essential oil as a primary outcome measure and have a regular menstrual cycle will participate. A menstrual cycle calendar will be created for the participants
Premenstrual Syndrome Scale (PMSS): | 1 year
  Participants in the study will be asked to fill in this scale. Women with premenstrual syndrome will be included in the study. The total score is obtained from the sum of the scores from all sub-dimensions. A minimum of 44 points and a maximum of 220 points can be obtained from the scale. An increase in the score obtained from the scale indicates that the intensity of the symptoms increases. If the total scale score (220) on the PMS scale exceeds 50% (110), PMS is considered "present".

SECONDARY OUTCOMES:
Premenstrual Syndrome Scale (PMSS): | 1 year
  Participants in the study will be asked to complete this scale in the 1st, 2nd and 3rd menstrual cycles. Women with premenstrual syndrome will be included in the study. The total score is obtained from the sum of the scores from all sub-dimensions. A minimum of 44 points and a maximum of 220 points can be obtained from the scale. An increase in the score obtained from the scale indicates that the intensity of the symptoms increases. PMS is considered "present" if the total scale score (220) on the PMS scale exceeds 50% (110).
SF-36 Quality of Life Scale | 1 year
  Participants in the study will be asked to complete this scale in the 1st, 2nd and 3rd menstrual cycles. The scale consists of eight sub-dimensions: physical function, physical role limitations, emotional role limitations, vitality (life energy), social function, pain, and mental health. and general health perception. A separate score is obtained for each subscale. The SF-36 evaluates the positive as well as the negative aspects of health status. Sub-dimension scores range from 0 to 100. The scores are positive. Increasing score indicates better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: özlem karabulutlu, assoc.dr, Principal Investigator — kafkas univesity

IPD SHARING:
Plan to Share IPD: No